CLINICAL TRIAL: NCT04282850
Title: Ablation Versus Medical Management of Atrial Fibrillation in Heart Failure With Preserved Ejection fRaction and the Effects on Exercise Capacity (AMPERE)
Brief Title: Ablation Versus Medical Management of Atrial Fibrillation in HFpEF
Acronym: AMPERE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Biosense Webster, Inc. (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U23-02-4965
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Heart Failure With Normal Ejection Fraction
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 2:1 randomization to catheter ablation (PVI) or to medical management.
Who Masked: Outcomes Assessor
Masking Description: Serum biomarkers, atrial fibrillation burden, anatomical and functional echocardiographic parameters, and exercise capacity will all be measured and analyzed by study personnel blinded to the patient's intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Vein Isolation (PVI) Group (Experimental): Subjects randomized to this treatment arm will undergo atrial fibrillation ablation, and undergo routine post-procedural follow-up.
  Interventions: Procedure: Pulmonary Vein Isolation
- Medical Management (No Intervention): Subjects randomized to this treatment arm will undergo medical management of the arrhythmia, but will not undergo invasive electrophysiologic procedures to address subject's AF.

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation — The intervention will involve standard of care electrophysiology ablation for rhythm management of atrial fibrillation with a procedure called a pulmonary vein isolation.
  Other Names: Atrial fibrillation ablation
  Arms: Pulmonary Vein Isolation (PVI) Group

SUMMARY:
This is a prospective non-blinded randomized control pilot study comparing the effect of pulmonary vein isolation against medical management of atrial fibrillation in patients with Heart Failure with preserved Ejection Fraction (HFpEF).

DETAILED DESCRIPTION:
Recent studies using PVI for rhythm control in patients with heart failure with reduced ejection fraction (HFrEF) have shown improvement in systolic ejection fraction, exercise capacity, quality of life, and a significant reduction in all-cause mortality. The PVI procedure has been shown to be safe and comparably effective in treating Atrial Fibrillation (AF) in HFpEF patients, but no studies have yet demonstrated the effects of catheter ablation on exercise capacity or clinical outcomes.

The investigators propose a prospective, non-blinded randomized control pilot study to assess the feasibility of conducting larger scale studies to determine if there are differences between catheter ablation with medical management on exercise capacity and quality of life in HFpEF patients with AF. The investigators' study will be powered for AF burden reduction, and the investigators hope to use the effect size on exercise capacity and heart failure events to help determine power for larger clinical studies that will follow to shed light on how invasive management of atrial fibrillation may impact the natural history of individuals with these two cardiovascular conditions.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 90 years of age, male or female
* Left Ventricular Ejection Fraction (LVEF) > 50% by echocardiogram during routine screening or within 12 months prior to enrollment day.
* Symptoms of heart failure requiring treatment with diuretic therapy for at least 30 days preceding enrollment.
* Symptomatic paroxysmal or persistent atrial fibrillation.
* Paroxysmal atrial fibrillation defined as recurrent AF (at least 2 episodes) that terminated spontaneously within 7 days
* Persistent AF was defined as AF which is sustained beyond 7 days, or lasting less than 7 days but necessitating pharmacologic or electrical cardioversion
* Included within the category of persistent AF is "long-standing persistent AF" defined as continuous AF of greater than 1 year in duration
* AF episodes had to be documented in the last 3 months prior to enrollment by ECG, Holter monitor, Loop recorder, memory of the implanted device, or any suitable device.
* Current symptoms of heart failure (NYHA II-IV) at the enrollment visit (Visit 1)
* Structural heart disease evidenced by one or both of the following echocardiographic findings (done during the transthoracic echocardiography (TTE) within 6 months of enrollment)
* Left atrial enlargement (LAE) defined as LA width > 3.8 cm or LA length > 5.0 cm, or LA area > 20 cm2 or LA volume > 55 mL or LA volume index > 29 ml/m2. (of note, LA length greater than 6.0 cm will be excluded)
* Left ventricular hypertrophy (LVH) defined by septal thickness or posterior wall thickness > 1.0 cm
* And at least one of the following:
* A heart failure hospitalization lasting over 12 hours and including intravenous diuretics at a healthcare facility within 12 months prior to the enrollment visit.
* An elevated pro-brain natriuretic peptide (BNP) (>100 pg/mL, or N-terminal pro b-type natriuretic peptide (NT-proBNP)>300 pg/mL)
* Hemodynamic testing consistent with HFpEF physiology including pulmonary capillary wedge pressure (PCWP) (or LVEDP) ≥ 15 mmHg.

Exclusion Criteria:

* Previous left heart ablation procedure for AF
* Contraindication to chronic anticoagulation therapy or heparin
* Longstanding atrial fibrillation, defined here as greater than 3 years of persistent atrial fibrillation
* Severe left atrial dilatation, with LA length > 6.0 cm, optimally from parasternal long view
* Acute coronary syndrome within 4 weeks as defined by electrocardiographic (ECG) ST segment depression or prominent T-wave inversion and/or positive biomarkers of necrosis (e.g. troponin) in the absence of ST-segment elevation and in an appropriate clinical setting (chest discomfort or angina equivalent).
* Cardiac surgery, angioplasty, or cerebrovascular accident within 4 weeks prior to enrollment.
* Planned cardiovascular intervention
* Listed for heart transplant
* Cardiac assist device implanted or need for mechanical hemodynamic support or inpatient admission
* Life expectancy less than 1 year
* Uncontrolled hypertension, defined as resting systolic blood pressure >190 and/or resting diastolic pressure>110
* Chronic Kidney Disease (CKD) stage 4-5 (GFR<25 ml/min/1.73m2), or on hemodialysis
* Cardiac diagnosis in addition to or other than HFpEF:
* Active myocarditis
* Hypertrophic obstructive cardiomyopathy
* Severe valvular disease
* Restrictive or constrictive cardiomyopathy, including known amyloidosis, sarcoidosis, hemochromatosis
* Complex congenital heart disease
* Constrictive pericarditis
* Severe pulmonary hypertension (RVSP > 60 mmHg), not secondary to HFpEF
* Non-cardiac pulmonary edema
* Clinical evidence of digoxin toxicity
* Sepsis
* Inability to comply with planned study procedures
* Pregnancy or nursing mothers
* Uncontrolled hypothyroidism or hyperthyroidism
* BMI of >65 kg/m2

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in AF burden as assessed by difference in percentage of time an individual is in AF | 3, 6, 9, and 12 months from intervention
  AF burden, described as the percentage of time an individual is in AF relative to the total amount of time analyzed. This outcome will be assessed at multiple intervals following intervention arm, using a continuous, implantable heart rhythm monitor. The investigators' focus will be on the change between pre-intervention AF burden and AF burden at 6 month follow-up.

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  All deaths within 12 months of the intervention arm.
Number of cardiovascular mortalities | 12 months
  The number of deaths attributable to cardiovascular causes occurring within 12 months of the intervention arm
Number of all-cause hospitalizations | 12 months
  The total number of inpatient hospitalizations within 12 months following the intervention.
Number of heart failure hospitalizations | 12 months
  The total number of inpatient hospitalizations attributable to heart failure exacerbations within 12 months following the intervention.
Change in patient-reported quality of life as assessed by Kansas City Cardiomyopathy Questionnaire | At enrollment (baseline) and 6 months following intervention
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. A change of 10 points or more is considered not only clinically significant but also carries prognostic implications for event-free survival in heart failure patients.
Change in NT pro-BNP levels | At enrollment (baseline) and 6 months following intervention
  Serum biomarker associated with congestive heart failure symptoms, measured in (mg/ml).
Change in exercise capacity as assessed by the 6 minute walk distance test | At baseline and 6 months post intervention
  Pre-intervention arm and 6 month post-procedural exercise capacity will be assessed using change in 6 minute walk distance, defined as the total distance (in meters) traversed during 6 minutes of time. This is well-validated measure of functional capacity and prognostic marker in patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Atwater, MD, Study Chair — Inova Heart and Vascular Institute; Eunice Yang, MD PhD, Principal Investigator — Inova Heart and Vascular Institute
Locations (1):
- Inova Heart and Vascular Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No